CLINICAL TRIAL: NCT00563888
Title: Change of Neural Network Indicators Through Narrative Treatment of PTSD in Torture Victims
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Konstanz (Other)
Collaborators: German Research Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SOSS-B6; SOSS-B6
Record Dates: First submitted 2007-11-23; First posted 2007-11-26 (Estimated); Last update posted 2007-11-26 (Estimated); Status verified 2007-11

CONDITIONS: PTSD
Keywords: PTSD; torture survivors; Narrative Exposure Therapy; trauma-related memory processes; steady state visual evoked fields
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Narrative Exposure Therapy (NET)
  Interventions: Behavioral: NET
- B (No Intervention): Waitinglist Control Group

INTERVENTIONS:
Behavioral: NET — Narrative Exposure Therapy for traumatized survivors of organized violence
  Arms: A

SUMMARY:
Effective Treatment of PTSD involves talking about the traumatic event in detail.It is unclear how this process influences the sensory-specific trauma network (fear structure)in the traumatized person. The goal of the project is to test the hypothesis that treatment-facilitated recovery does not change the original fear structure but establishes an inhibitory mechanism that depends on verbal activity. An affective visual steady-state paradigm in magnetencephalography (MEG) using positive, aversive and neutral picture stimuli will be used to examine the spatial and temporal pattern of the processing of emotional stimuli. To examine the effects of treatment this paradigm will be used as outcome measure within a randomized controlled trial of Narrative Exposure Therapy and a waiting-list control condition for severely traumatized torture victims.

ELIGIBILITY:
Inclusion Criteria:

* experiences of organized violence/torture
* PTSD diagnosis

Exclusion Criteria:

* psychotic disorder
* neurological disease or seizures
* current drug/alcohol abuse

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2007-01; Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
PTSD diagnosis and severity score according to the Clinicians Administered PTSD Scale (CAPS) | 4 & 9 months after completion of treatment

SECONDARY OUTCOMES:
steady state visual evoked magnetic fields in response to affective stimuli | 4 & 9 months after completion of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Catani, Dr., Study Director — University of Konstanz; Frank Neuner, Prof., Principal Investigator — University of Konstanz
Locations (1):
- University of Konstanz, Department of Psychology, Konstanz, Germany

REFERENCES:
- [Derived] Adenauer H, Catani C, Gola H, Keil J, Ruf M, Schauer M, Neuner F. Narrative exposure therapy for PTSD increases top-down processing of aversive stimuli--evidence from a randomized controlled treatment trial. BMC Neurosci. 2011 Dec 19;12:127. doi: 10.1186/1471-2202-12-127. PMID 22182346
- [Derived] Adenauer H, Pinosch S, Catani C, Gola H, Keil J, Kissler J, Neuner F. Early processing of threat cues in posttraumatic stress disorder-evidence for a cortical vigilance-avoidance reaction. Biol Psychiatry. 2010 Sep 1;68(5):451-8. doi: 10.1016/j.biopsych.2010.05.015. PMID 20619396